CLINICAL TRIAL: NCT04866225
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE, 2-PERIOD STUDY IN HEALTHY ADULT MALE PARTICIPANTS TO ASSESS THE EXTENT OF EXCRETION, ABSOLUTE BIOAVAILABILITY, FRACTION ABSORBED, AND PHARMACOKINETICS OF [14C]PF-06865571 USING A 14C-MICROTRACER APPROACH
Brief Title: A Study in Healthy Adult Male Participants to Assess Absorption, Distribution, Metabolism and Excretion (ADME) of Radiolabeled PF-06865571.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C2541007
Record Dates: First submitted 2021-04-19; First posted 2021-04-29 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-02

CONDITIONS: Healthy Participants
Keywords: ADME
MeSH Terms: interventions — ervogastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): One arm of healthy male participants administered a single oral dose of [14C]PF-06865571; followed by a single dose of unlabeled PF-06865571, and IV administration of [14C]PF-06865571 three hours later.
  Interventions: Drug: Oral [14C]PF-06865571; Drug: Oral PF-06865571; Drug: IV [14C]PF-06865571

INTERVENTIONS:
Drug: Oral [14C]PF-06865571 — Oral radiolabeled PF-06865571
Drug: Oral PF-06865571 — Oral PF-06865571
Drug: IV [14C]PF-06865571 — IV radiolabeled PF-06865571

SUMMARY:
This study is a Phase 1, open-label, non-randomized, 2-period, fixed-sequence, single-dose study of PF-06865571 in healthy male participants to characterize the ADME properties of [14C]PF-06865571 following oral administration; and to evaluate the absolute oral bioavailability (F) and fraction absorbed (Fa) of PF-06865571 following oral administration of unlabeled PF-06865571 and IV administration of [14C]PF-06865571.

ELIGIBILITY:
Inclusion Criteria:

* Male participants, 18 to 60 years of age, inclusive, at the time of signing the informed consent document.
* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac tests.
* Participants who are nonsmoking for at least 3 months at the time of signing the informed consent document.
* BMI of 17.5 to 30.4 kg/m2, inclusive; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of irregular bowel movements including irritable bowel syndrome or frequent episodes of diarrhea or constipation, defined by less than 1 bowel movement on average per 2 days, or lactose intolerance.
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg,or HCVAb. Hepatitis B vaccination is allowed.
* History of SARS-CoV-2 PCR or antibody (eg, IgG, IgM, etc) positive result would necessitate accompanying history of asymptomatic state for at least 6 months prior to screening.
* Use of prescription or nonprescription drugs.
* Previous administration with an unapproved drug within 60 days preceding the first dose of study intervention used in this study.
* A positive urine drug test.
* A positive urine cotinine test.
* A positive COVID-19 (SARS-CoV-2) PCR test.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Labcorp Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2541007

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1:[14C]PF-06865571 300 mg Oral; Period 2:PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV: Six healthy male participants were enrolled and received 2 regimens (A and B) in Periods 1 and 2, respectively. For regimen A in Period 1, an oral dose of 300 mg PF-06865571 containing approximately 300 nCi 14C (ie, radiolabeled PF-06865571) was administered. For regimen B in Period 2, an oral dose of 300 mg unlabeled PF-06865571 followed by an intravenous (IV) dose of 300 nCi [14C] in 100 μg of PF-06865571 was administered.
Period: Overall Study
Arm/Group | Period 1:[14C]PF-06865571 300 mg Oral; Period 2:PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Arm/Group | Period 1:[14C]PF-06865571 300 mg Oral; Period 2:PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 42.0 (13.90)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-25 years | 1
  26-35 years | 1
  36-45 years | 1
  >45 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4
  Black or African American | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Recovery of Radioactivity in Urine as Percentage of Total Radioactive Dose of PF-06865571 Administered
Description: The total recovery of radioactivity in urine was listed and summarized using descriptive statistics. In this outcome measure, the percentages of dose excreted in urine in Period 1 and Period 2 were reported.
Time Frame: Period 1: Day -1 to maximum Day 21; Period 2: Day 1 to maximum Day 3
Population: Analysis population included all participants who received 1 dose of [14C]PF-06865571 and who have evaluable total radioactivity concentration (urinary and fecal) data and who had no protocol deviations or AEs (such as vomiting of the dose, diarrhoea or severe constipation) that may have affected the extent of excretion analysis.
Measure: Mean (Standard Deviation); unit: Percentage of Dose
Groups:
- [14C]PF-06865571 300 mg Oral: An oral single-dose of 300 mg PF-06865571 containing approximately 300 nCi 14C (ie, radiolabeled PF-06865571) was administered on Day 1 in Period 1.
- PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV: An oral single-dose of 300 mg unlabeled PF-06865571 followed by an IV dose of 300 nCi [14C] in 100 μg of PF-06865571 (at around 3 hours post oral dose) was administered on Day 1 in Period 2. The [14C] IV dose was administered as an infusion over approximately 15 minutes.
Arm/Group | [14C]PF-06865571 300 mg Oral | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6 | 6
Percentage of Dose | 48.9 (16.3) | 51.5 (15.8)

2. Primary Outcome: Total Recovery of Radioactivity in Feces as Percentage of Total Radioactive Dose of PF-06865571 Administered
Description: The total recovery of radioactivity in feces was listed and summarized using descriptive statistics. In this outcome measure, the percentages of dose excreted in feces in Period 1 and Period 2 were reported.
Time Frame: Period 1: Day -1 to maximum Day 21; Period 2: Day 1 to maximum Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Dose
Arm/Group | [14C]PF-06865571 300 mg Oral | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6 | 6
Percentage of Dose | 30.1 (2.9) | 18.8 (3.3)

3. Primary Outcome: Total Recovery of Radioactivity in Total Excreta (Urine + Feces) as Percentage of Total Radioactive Dose of PF-06865571 Administered
Description: The total recovery of radioactivity in the combination of urine and feces was listed and summarized using descriptive statistics. In this outcome measure, the percentages of dose excreted in total excreta (urine + feces) in Period 1 and Period 2 were reported.
Time Frame: Period 1: Day -1 to maximum Day 21; Period 2: Day 1 to maximum Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Dose
Arm/Group | [14C]PF-06865571 300 mg Oral | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6 | 6
Percentage of Dose | 79.0 (16.7) | 70.3 (15.1)

4. Primary Outcome: Relative Abundance (Mean Value) of Radiolabeled PF-06865571 in Plasma in Period 1
Description: Plasma samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in plasma, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of radiolabeled PF-06865571 in plasma based on [14C] quantitation was reported. The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Number; unit: Percentage of Radioactivity in Plasma
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Plasma | 43.8

5. Primary Outcome: Relative Abundance (Mean Value) of Metabolites of Radiolabeled PF-06865571 in Plasma in Period 1
Description: Plasma samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in plasma, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of the metabolites of [14C]PF-06865571 in plasma based on [14C] quantitation was reported. The metabolites included 487, 391, 412, 556, M6 (PF-07822633), M7 (PF-07911964), 584, M1 (PF-06878236), 426, M4 (PF-06887477), 600, M5 (PF-06885984) and M2 (PF-06868609). The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: 0, 0.5, 3, 6, 12, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: as for outcome 4
Measure: Number; unit: Percentage of Radioactivity in Plasma
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Plasma
  487 | 0
  391 | 3.0
  412 | 0
  556 | 2.7
  M6 (PF-07822633) | 11.3
  M7 (PF-07911964) | 0.01
  584 | 1.1
  M1 (PF-06878236) | 0
  426 | 1.5
  M4 (PF-06887477) | 1.5
  600 | 0
  M5 (PF-06885984) | 0
  M2 (PF-06868609) | 36.6

6. Primary Outcome: Relative Abundance (Mean Value) of Radiolabeled PF-06865571 in Urine in Period 1
Description: Urine samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in urine, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of radiolabeled PF-06865571 in urine based on [14C] quantitation was reported. The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: Day -1 to maximum Day 21
Population: as for outcome 4
Measure: Number; unit: Percentage of Radioactivity in Urine
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Urine | 2.7

7. Primary Outcome: Relative Abundance (Mean Value) of Metabolites of Radiolabeled PF-06865571 in Urine in Period 1
Description: Urine samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in urine, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of the metabolites of [14C]PF-06865571 in urine based on [14C] quantitation was reported. The metabolites included 487, 391, 412, 556, M6 (PF-07822633), M7 (PF-07911964), 584, M1 (PF-06878236), 426, M4 (PF-06887477), 600, M5 (PF-06885984) and M2 (PF-06868609). The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: Day -1 to maximum Day 21
Population: as for outcome 4
Measure: Number; unit: Percentage of Radioactivity in Urine
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Urine
  487 | 2.0
  391 | 6.0
  412 | 0
  556 | 4.7
  M6 (PF-07822633) | 23.3
  M7 (PF-07911964) | 23.3
  584 | 23.3
  M1 (PF-06878236) | 0.7
  426 | 4.2
  M4 (PF-06887477) | 4.2
  600 | 1.4
  M5 (PF-06885984) | 1.4
  M2 (PF-06868609) | 50.9

8. Primary Outcome: Relative Abundance (Mean Value) of Radiolabeled PF-06865571 in Feces in Period 1
Description: Fecal samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in feces, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of radiolabeled PF-06865571 in feces based on [14C] quantitation was reported. The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: Day -1 to maximum Day 21
Population: as for outcome 4
Measure: Number; unit: Percentage of Radioactivity in Feces
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Feces | 4.1

9. Primary Outcome: Relative Abundance (Mean Value) of Metabolites of Radiolabeled PF-06865571 in Feces in Period 1
Description: Fecal samples were analyzed for radiolabeled PF-06865571 and its metabolites. [14C]PF-06865571 and the major metabolites in feces, after oral administration of 300 mg [14C]PF-06865571 were identified. In this outcome measure, relative abundance of the metabolites of [14C]PF-06865571 in feces based on [14C] quantitation was reported. The metabolites included 487, 391, 412, 556, M6 (PF-07822633), M7 (PF-07911964), 584, M1 (PF-06878236), 426, M4 (PF-06887477), 600, M5 (PF-06885984) and M2 (PF-06868609). The measure type was the mean value based on pooled sampling, which means blood samples from the 6 participants were pooled together and then analyzed as 1 sample, thus the confidence interval could not be calculated. Therefore, "Number" is selected as the Measure Type.
Time Frame: Period 1: Day -1 to maximum Day 21
Population: as for outcome 4
Measure: Number; unit: Percentage of Radioactivity in Feces
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Radioactivity in Feces
  487 | 0
  391 | 0
  412 | 1.1
  556 | 0
  M6 (PF-07822633) | 0
  M7 (PF-07911964) | 21.0
  584 | 0
  M1 (PF-06878236) | 15.0
  426 | 33.2
  M4 (PF-06887477) | 33.2
  600 | 0
  M5 (PF-06885984) | 0
  M2 (PF-06868609) | 23.1

10. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time Zero to Time of The Last Quantifiable Concentration (AUClast) of Total Radioactivity of [14C]PF-06865571 in Plasma in Period 1
Description: AUClast is defined as area under the plasma concentration-time profile from time zero to time of the last quantifiable concentration (Clast). The determination method of AUClast was linear/log trapezoidal rule.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL (ngEq = nanogram equivalent)
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ngEq*hr/mL (ngEq = nanogram equivalent) | 20080 (15)

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Total Radioactivity of [14C]PF-06865571 in Plasma in Period 1
Description: Cmax is defined as maximum plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL (nanogram-equivalent/milliliter)
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ngEq/mL (nanogram-equivalent/milliliter) | 4417 (10)

12. Secondary Outcome: Time for Cmax (Tmax) of Total Radioactivity of [14C]PF-06865571 in Plasma in Period 1
Description: Tmax is defined as time to reach maximum observed plasma concentration. The determination method of Tmax was observing directly from data as time of first occurrence.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Median (Full Range); unit: hr (hours)
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
hr (hours) | 3.00 [3.00 to 4.00]

13. Secondary Outcome: Area Under the Plasma Concentration Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Total Radioactivity of [14C]PF-06865571 in Plasma in Period 1
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). The determination method of AUCinf was AUClast + (Clast*/ kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, kel was the terminal phase rate constant.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ngEq*hr/mL | 20400 (15)

14. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Total Radioactivity of [14C]PF-06865571 in Plasma in Period 1
Description: Terminal elimination half-life (t1/2) was the time measured for the plasma concentration to decrease by one half. The determination method of t1/2 was loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
hr | 3.622 (1.9605)

15. Secondary Outcome: AUClast of Oral PF-06865571 in Plasma in Period 1
Description: as for outcome 10
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL (nanogram*hour per milliliter)
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ng*hr/mL (nanogram*hour per milliliter) | 7962 (19)

16. Secondary Outcome: Cmax of Oral PF-06865571 in Plasma in Period 1
Description: Cmax is defined as maximum plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL (nanogram per milliliter)
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ng/mL (nanogram per milliliter) | 2096 (15)

17. Secondary Outcome: Tmax of Oral PF-06865571 in Plasma in Period 1
Description: as for outcome 12
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
hr | 3.00 [2.00 to 4.00]

18. Secondary Outcome: AUCinf of Oral PF-06865571 in Plasma in Period 1
Description: as for outcome 13
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
ng*hr/mL | 7964 (19)

19. Secondary Outcome: t1/2 of Oral PF-06865571 in Plasma in Period 1
Description: as for outcome 14
Time Frame: Period 1: 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose (Day 1 to Day 6)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
hr | 6.275 (2.9246)

20. Secondary Outcome: AUClast of Intravenous (IV) Radiolabeled PF-06865571 in Plasma in Period 2
Description: as for outcome 10
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
ng*hr/mL | 4.145 (20)

21. Secondary Outcome: Cmax of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: Cmax is defined as maximum plasma concentration. The determination method of Cmax was observing directly from data.
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
ng/mL | 2.893 (13)

22. Secondary Outcome: Tmax of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: as for outcome 12
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
hr | 0.250 [0.167 to 0.250]

23. Secondary Outcome: t1/2 of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: as for outcome 14
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
hr | 1.232 (0.25664)

24. Secondary Outcome: AUCinf of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: as for outcome 13
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
ng*hr/mL | 4.209 (19)

25. Secondary Outcome: Systemic Clearance (CL) of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. The determination method of CL was dose/AUCinf.
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr (liter per hour)
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
L/hr (liter per hour) | 23.88 (20)

26. Secondary Outcome: Steady State Volume of Distribution (Vss) of IV Radiolabeled PF-06865571 in Plasma in Period 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L (Liters)
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
L (Liters) | 38.83 (16)

27. Secondary Outcome: Dose-Normalized AUCinf (AUCinf[dn]) of Oral Unlabeled PF-06865571 in Plasma in Period 2
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf). AUCinf(dn) is defined as dose normalized (to 1 mg equivalent) AUCinf, which equals to AUCinf/Dose.
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
ng*hr/mL/mg | 31.46 (21)

28. Secondary Outcome: AUCinf(dn) of IV Microtracer of Radiolabeled PF-06865571 in Plasma in Period 2
Description: as for outcome 27
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
ng*hr/mL/mg | 41.92 (20)

29. Secondary Outcome: Absolute Oral Bioavailability (F) of Oral Unlabeled and IV Radiolabeled PF-06865571 for Plasma AUCinf(dn) in Period 2
Description: Absolute Oral Bioavailability (F) provided information on the amount of PF-06865571 reaching the systemic circulation. F was estimated as the ratio of adjusted geometric means of dose-normalized AUCinf for oral unlabeled PF-06865571 and IV labeled 14C PF-06865571 in plasma (from Period 2 only) which was equivalent to the following equation: F = [PF-06865571_AUCpo/[14C]PF-06865571_AUCiv]×[ [14C]PF-06865571_Doseiv/ PF-06865571_Dosepo], where PF-06865571_AUCpo = AUCinf(dn) of oral unlabeled PF-06865571, [14C]PF-06865571_AUCiv = AUCinf(dn) of intravenous radiolabeled PF-06865571, [14C]PF-06865571_Doseiv = dose of intravenous radiolabeled PF-06865571, PF-06865571_Dosepo = dose of oral unlabeled PF-06865571.
Time Frame: Period 2: -3, 0, 0.08, 0.17, 0.25, 0.5, 0.75, 1, 3, 6, 9, 13, 21, 33 and 45 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the PF-06895571 PK parameters of interest and at least one of the 14C parameters of interest.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
Percent | 75.06 [71.06 to 79.29]

30. Secondary Outcome: Percentage of Total 14C in Urine Following Oral Administration (%14C_Urine_PO) of Radiolabeled PF-06865571 in Period 1
Description: %14C_Urine_PO is defined as percentage of the radioactive dose administered that is excreted in the urine following oral administration. %14C_Urine_PO = Total 14C_Urine_PO/14C Dosepo × 100, where PO = orally, Total 14C_Urine_PO = total radioactivity excreted into the urine post-dose following oral administration of [14C]PF-06865571, 14C Dosepo = dose of 14C following oral administration of [14C]PF-06865571.
Time Frame: Period 1: up to 48 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Total 14C
Arm/Group | [14C]PF-06865571 300 mg Oral
Number analyzed (Participants) | 6
Percentage of Total 14C | 45.92 (44)

31. Secondary Outcome: Percentage of Total 14C in Urine Following IV Microtracer Administration (%14C_Urine_IV) of Radiolabeled PF-06865571 in Period 2
Description: %14C_Urine_IV is defined as percentage of the radioactive dose administered that is excreted in the urine following IV administration. %14C_Urine_IV = Total 14C _Urine_IV/14C Doseiv × 100, where IV = intravenous, Total 14C_Urine_IV = total radioactivity excreted into the urine following IV administration of [14C]PF 06865571, 14C Doseiv = dose of 14C following IV administration of [14C]PF 06865571.
Time Frame: Period 2: up to 48 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Total 14C
Arm/Group | PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
Percentage of Total 14C | 49.50 (44)

32. Secondary Outcome: Fraction Absorbed (Fa) for Percentage of Excretion of Total 14C in Urine for Oral and IV Radiolabeled PF-06865571
Description: Determination of the Fraction Absorbed (Fa) (obtained from Periods 1 and 2) provided information on the fraction of the total PF-06865571 dose absorbed, regardless of the fate of that dose after absorption (ie, metabolism, degradation, etc). Fa was estimated as the ratio of the adjusted geometric means of % of administered radioactive dose excreted into the urine following oral and IV administration of [14C]PF-06865571 microtracer dose over the same collection time (up to 48 hours post dose) in Periods 1 and 2, respectively: Fa = [% 14C_Urine_PO/% 14C_Urine_IV].
Time Frame: Period 1 and Period 2: up to 48 hours post-dose (Day 1 to Day 3)
Population: Analysis population included all participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (90% Confidence Interval); unit: Percent
Groups:
- [14C]PF-06865571 300 mg Oral; PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV: [14C]PF-06865571 300 mg oral: an oral single-dose of 300 mg PF-06865571 containing approximately 300 nCi 14C (ie, radiolabeled PF-06865571) was administered on Day 1 in Period 1.
  PF-06865571 300 mg oral & [14C]PF-06865571 100 μg IV: an oral single-dose of 300 mg unlabeled PF-06865571 followed by an IV dose of 300 nCi [14C] in 100 μg of PF-06865571 (at around 3 hours post oral dose) was administered on Day 1 in Period 2. The [14C] IV dose was administered as an infusion over approximately 15 minutes.
Arm/Group | [14C]PF-06865571 300 mg Oral; PF-06865571 300 mg Oral & [14C]PF-06865571 100 μg IV
Number analyzed (Participants) | 6
Percent | 92.78 [62.07 to 138.68]

ADVERSE EVENTS:
Time Frame: For Period 1, adverse events were assessed from Baseline up to Day 21. For Period 2, adverse events were assessed from Baseline up to Day 21, followed by one follow-up phone call for each participant which occurred at least 28 days and up to 35 days after the last dose of PF-06865571.
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- [14C] PF-06865571 300 mg Oral: An oral single-dose of 300 mg PF-06865571 containing approximately 300 nCi 14C (ie, radiolabeled PF-06865571) was administered on Day 1 in Period 1.
- PF-06865571 300 mg Oral & [14C] PF-06865571 100 μg IV: An oral single-dose of 300 mg unlabeled PF-06865571 followed by an IV dose of 300 nCi [14C] in 100 μg of PF-06865571 (at around 3 hours post oral dose) was administered on Day 1 in Period 2. The [14C] IV dose was administered as an infusion over approximately 15 minutes.
Arm/Group | [14C] PF-06865571 300 mg Oral | PF-06865571 300 mg Oral & [14C] PF-06865571 100 μg IV
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | [14C] PF-06865571 300 mg Oral (N=6) | PF-06865571 300 mg Oral & [14C] PF-06865571 100 μg IV (N=6)
Conjunctivitis allergic (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04866225/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04866225/SAP_001.pdf